CLINICAL TRIAL: NCT01814124
Title: Therapeutic Effectiveness of Manual Therapy Plus Exercise for Femoroacetabular Impingement of the Hip: a Randomized Controlled Clinical Trial Pilot Study
Brief Title: Conservative Management of Femoroacetabular Impingement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: High Point University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201207-116
Record Dates: First submitted 2013-03-14; First posted 2013-03-19 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Femoroacetabular Impingement
MeSH Terms: conditions — Femoracetabular Impingement | interventions — Musculoskeletal Manipulations; Exercise; Counseling

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Advice and home exercise (Active Comparator): All participants will be given a handout consisting of education about avoidance of certain activities as well as 3 stretches and 3 strengthening exercises to be performed as a home exercise program 2-3x/week
  Interventions: Other: Advice and home exercise
- Manual Therapy Plus Exercise (Experimental): Participants in this group will be given the same handout consisting of education about avoidance of certain activities as well as 3 stretches and 3 strengthening exercises to be performed as a home exercise program 2-3x/week.
  Participants in this group will also receive 12 individualized physical therapy treatment sessions (2x/week for 6 weeks) consisting of both manual therapy and exercise directed at the hip and surrounding areas based upon findings from the initial examination. Participants will also be given additional exercises to be performed at home as directed by the treating physical therapist
  Interventions: Other: Manual therapy plus exercise; Other: Advice and home exercise

INTERVENTIONS:
Other: Manual therapy plus exercise
  Arms: Manual Therapy Plus Exercise
Other: Advice and home exercise

SUMMARY:
Femoroacetabular impingement (FAI) is recognized as a formal source of hip pain and disability typically affecting the young adult, active population and has been identified as a precursor to hip osteoarthritis (OA). Common impairments include sharp, anterior groin pain in a position of hip flexion limiting patients' ability to tolerate prolonged sitting, squatting, stair climbing, etc. resulting in both work limitations and decreased social participation. Manual therapy and exercise is known to be effective in reducing pain and increasing physical function in the management of hip OA. To the extent that FAI is often a precursor to developing hip OA, logic would seem to dictate a manual therapy plus exercise approach to decrease pain and disability and potentially prevent or delay osteoarthritis related surgery. Currently, surgery is considered the first line of treatment with respect to FAI. However, there is a lack of evidence to support or refute the use of conservative treatment interventions in this patient population.

This study is designed to investigate the benefits of physical therapy interventions (manual therapy and exercise) over usual care for improving pain and physical function in patients with FAI of the hip. For this study, 52 participants will be recruited from the Department of Orthopaedic Surgery, Wake Forest Baptist Medical Center, for an outpatient consultation for consideration of hip arthroscopy surgery. Participants will include those patients who meet clinical and radiological criteria for formal diagnosis of FAI. Participants will be randomized into two treatment groups. Participants in one group will receive usual care plus manual therapy directed at the hip as well as a supervised exercise program and home exercise program twice weekly for six weeks. Participants in the usual care group will receive usual care as prescribed by the physician. Changes in pain, physical function and benefits of the intervention will be assessed over six weeks. Should this research study demonstrate treatment effectiveness of physical therapy intervention in patients diagnosed with FAI of the hip, manual therapy plus exercise may have the potential to delay or prevent surgery in this patient population. Further, to the extent to which FAI has been shown to lead to later development of hip OA, effective treatment interventions may help to delay or prevent secondary osteoarthritis related changes as well as total joint replacement surgery associated with hip OA. This study will provide preliminary data that can be used to prepare further grant applications designed to determine the safest, most effective treatments for patients with FAI.

ELIGIBILITY:
Inclusion Criteria:

* The participants will include new and existing patients with a diagnosis of femoroacetabular impingement and are being seen for an outpatient consultation for consideration of hip arthroscopy surgery.
* From direct correspondence with Dr. Stubbs, criteria for formal diagnosis of FAI includes a combination of clinical diagnosis supported with radiography.
* Clinical examination typically consists of reported hip pain, decreased flexion (<95o), decreased internal rotation (<10o), and
* a positive anterior impingement test result (report of deep, anterior groin pain following combination of flexion, internal rotation, and adduction).
* Use of an alpha angle is also used as a distinct characteristic with patient's having an alpha angle of > 50-55 degrees at increased risk for FAI.

Exclusion Criteria:

* previous hip surgery;
* any other surgical procedure of the lower limbs in the prior 6 months;
* pre-existing disease state of the hip such as rheumatoid arthritis;
* fracture;
* congenital/developmental hip dysplasia;
* initiation of opioid analgesia or cortico-steroid or analgesic injection intervention for hip pain within prior 30 days;
* physical impairments unrelated to the hip preventing safe participation in exercise, manual therapy, walking or stationary cycling;
* advanced osteoporosis;
* body mass index > 38;
* significant cardio-pulmonary disease;
* cardiac pacemaker;
* stated inability to complete the proposed course of intervention and follow-up;
* insufficient English language skills to comprehend assessment tools;
* resident greater than 90 minutes from Wake Forest Baptist Medical Center.
* Individuals with contraindications to treatment with mobilization and manipulation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2013-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Hip Outcome Score | Change from baseline functional status at 6 weeks
  Participants will fill out the Hip Outcome Score (HOS). The HOS is a 29-item instrument. Patient data from the HOS has been reported as reliable, valid, and responsive specific to this patient population and has been identified as the best available questionnaire for assessing younger patients undergoing hip arthroscopy. Test-retest reliability has been reported in the range of ICC = 0.92 - 0.98; internal consistency measures at cronbach's alpha = 0.96, 0.95; and responsiveness characteristics with effect sizes post-surgery ranging from 1.2-1.5.
Numeric Pain Rating Scale | Change from baseline pain level at 6 weeks
  Lower extremity pain will be recorded using the Numeric Pain Rating Scale (NPRS). Participants will be asked to report their pain levels from no pain (0/10) to worse imaginable pain (10/10). This scale has been demonstrated to be a reliable, generalizable, internally consistent measure of clinical and experimental pain sensation intensity.

SECONDARY OUTCOMES:
Functional Squat | Change from baseline functional status at 6 weeks
  The functional squat test is considered to be a provocative test that also serves as a measure of function. A digital inclinometer will be placed on the tibia just distal to the tibial tuberosity. The participants will be asked to bend the knees and bring their buttocks toward their heels without bending forward or lifting their heels off the floor. The range of motion measurement will be taken at the greatest range of motion at which the participant was able to maintain good form or the first point of reported pain. The functional squat test has good reported reliability (ICC = 0.90 - 0.92) and responsiveness with standard error of measurement of 1.9.
Global Rating of Change Scale | 6 weeks
  The Global Rating of Change Scale (GRCS) will be completed by each participant to rate their own perception of improved hip function. The GRCS questionnaire is an instrument that measures overall changes in the quality of life of the subject. The use of a GRCS is a common, feasible, and useful method for assessing outcome, and has been shown to be a valid measurement of change in patient status in patients with knee OA and other pain populations
Lower Extremity Functional Scale | Change from baseline general functional status at 6 weeks
  General lower extremity function will be quantified using the LEFS. The LEFS is a 20 item instrument with reported test-retest reliability of ICC = 0.98; internal consistency measures of cronbach's alpha = 0.96; and responsiveness characteristics of area under the curve of 0.77

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Human Health and Sports Science Research, High Point, North Carolina, United States

REFERENCES:
- [Derived] Wright AA, Hegedus EJ, Taylor JB, Dischiavi SL, Stubbs AJ. Non-operative management of femoroacetabular impingement: A prospective, randomized controlled clinical trial pilot study. J Sci Med Sport. 2016 Sep;19(9):716-21. doi: 10.1016/j.jsams.2015.11.008. Epub 2016 Jan 6. PMID 26795448